CLINICAL TRIAL: NCT05712902
Title: A Phase II, Single Arm, Multicenter Study to Evaluate Anti-tumor Activity, Safety, Tolerability and Pharmacokinetics of DZD9008 in Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) with EGFR Exon 20 Insertion Mutation
Brief Title: Sunvozertinib (DZD9008) in Pretreated Lung Cancer Patients with EGFR Exon20 Insertion Mutation (WU-KONG6)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2020E0001
Record Dates: First submitted 2023-01-12; First posted 2023-02-06 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daily dose of Sunvozertinib (Experimental)
  Interventions: Drug: Sunvozertinib

INTERVENTIONS:
Drug: Sunvozertinib — Daily dose of Sunvozertinib
  Other Names: DZD9008

SUMMARY:
This is a Phase II, single-arm, multi-center clinical study to evaluate the anti-tumor efficacy, safety, tolerability and pharmacokinetics of Sunvozertinib in participants with locally advanced or metastatic NSCLC carrying EGFR exon 20 insertion mutations whose disease has progressed on prior platinum-based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand the nature of the trial and provide a signed and dated, written informed consent form.
2. Aged at least 18 years old.
3. Histological or cytological confirmed locally advanced or metastatic NSCLC
4. Tumor tissue EGFR exon 20 insertion mutations confirmed by qualified local laboratories or sponsor-designated central laboratories.
5. Participants must exhibit Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1 at ICF signature with no deterioration over the past 2 weeks.
6. Predicted life expectancy ≥ 12 weeks.
7. Patient must have measurable disease according to RECIST 1.1.
8. Patients with brain metastasis (BM) can only be enrolled under the condition that BM is previously treated and stable.
9. Adequate organ system functions.
10. Patients should receive at least one line but no more than three lines of prior systemic therapy (at least one line must contain platinum-based therapy).

Exclusion Criteria:

1. Prior malignancy within 2 years requires active treatment, except for adequately treated basal cell skin carcinoma, in situ cervical carcinoma, or other cancer types (to be discussed with Dizal's Study Physician) who has been disease free for > 2 years with life expectancy >2 years.
2. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting Sunvozertinib with the exception of alopecia and grade 2 prior platinum-therapy related neuropathy.
3. Spinal cord compression or leptomeningeal metastasis.
4. History of stroke or intracranial hemorrhage within 6 months before first administration of Sunvozertinib.
5. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses.
6. Active infection including hepatitis B, hepatitis C, human immunodeficiency virus (HIV) and COVID-19.
7. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs).
   * Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, third degree heart block, and second-degree heart block, PR interval > 250 msec.
   * Any factors that increase the risk of QTc prolongation, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval .
   * Prior history of atrial fibrillation within 6 months of first administration of Sunvozertinib, except prior drug treatment related and recovered.
8. Participants with hemorrhagic diseases such as von Willebrand disease.
9. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease or immunotherapy induced immune pneumonia.
10. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of Sunvozertinib.
11. Prior/concomitant therapy

    1. Patients who have received prior Poziotinib, TAK-788, CLN-081 or BDTX-189, furmonertinib or any other EGFR/HER2 exon20ins small molecule inhibitors treatment should be excluded.
    2. Other EGFR TKIs, such as gefitinib, erlotinib, osimertinib, afatinib, dacomitinb are not considered EGFR or HER2 Exon20ins small molecule inhibitors, and thus prior treatment with these drugs is allowed unless the patient had an objective response and subsequent progression as assessed by the investigator or treating physician during treatment with that prior TKI.
    3. Treatment with antibodies within 4 weeks before first administration of Sunvozertinib.
    4. Any cytotoxic chemotherapy, investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days before first administration of Sunvozertinib.
12. Women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) according to RECIST 1.1 by an Independent Review Committee (IRC) | From first dosing until disease progression or intolerable adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, Principal Investigator — Peking Union Medical College Hospital
Locations (33):
- China (33):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital，Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital(The Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Army Medical Center of PLA, Chongqing
  - Chongqing University Cancer Hospital(Chongqing Cancer Hospital), Chongqing
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Hainan General Hospital, Haikou
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital (Cancer Hospital of the University of Chinese Academy of Sciences), Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The Second Hospital of Anhui Medical University, Hefei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Jinan Central Hospital (Central Hospital Affiliated to Shandong First Medical University), Jinan
  - Yunnan Cancer Hospital, Kunming
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Fudan University Shanghai Cancer Center, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi
  - Hubei Cancer Hospital, Wuhan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Affiliated Cancer Hospital of Zhengzhou University(Henan Cancer Hospital), Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang M, Fan Y, Sun M, Wang Y, Zhao Y, Jin B, Hu Y, Han Z, Song X, Liu A, Tang K, Ding C, Liang L, Wu L, Gao J, Wang J, Cheng Y, Zhou J, He Y, Dong X, Yao Y, Yu Y, Wang H, Sun S, Huang J, Fang J, Li W, Wang L, Ren X, Zhou C, Hu Y, Zhao D, Yang R, Xu F, Huang Y, Pan Y, Cui J, Xu Y, Yang Z, Shi Y. Sunvozertinib for patients in China with platinum-pretreated locally advanced or metastatic non-small-cell lung cancer and EGFR exon 20 insertion mutation (WU-KONG6): single-arm, open-label, multicentre, phase 2 trial. Lancet Respir Med. 2024 Mar;12(3):217-224. doi: 10.1016/S2213-2600(23)00379-X. Epub 2023 Dec 12. PMID 38101437